CLINICAL TRIAL: NCT04956640
Title: A Phase 1/2 Study of LY3537982 in Patients With KRAS G12C-Mutant Advanced Solid Tumors
Brief Title: Study of LY3537982 in Cancer Patients With a Specific Genetic Mutation (KRAS G12C)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LOXO-RAS-20001; 2021-000595-12 (EudraCT Number); J3M-OX-JZQA (Other: Eli Lilly and Company); MK-3475-E27/KEYNOTE E27 (Other: Merck Sharp & Dohme LLC); 2022-502756-31-00 (EU CTIS Number)
Record Dates: First submitted 2021-07-02; First posted 2021-07-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms
Keywords: Frontline; 1L; First Line
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — pembrolizumab; Cetuximab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3537982 (Dose Escalation) (Experimental): LY3537982 administered orally.
  Interventions: Drug: LY3537982
- LY3537982 (Dose Expansion) (Experimental): LY3537982 administered orally either alone or with another investigational agent.
  Interventions: Drug: LY3537982; Drug: Pembrolizumab; Drug: Cetuximab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- LY3537982 (Dose Optimization) (Experimental): LY3537982 administered orally either alone or with another investigational agent
  Interventions: Drug: LY3537982; Drug: Pembrolizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: LY3537982 — Oral
  Other Names: Olomorasib
Drug: Pembrolizumab — Intravenous
  Other Names: KEYTRUDA®
  Arms: LY3537982 (Dose Expansion); LY3537982 (Dose Optimization)
Drug: Cetuximab — Intravenous
  Other Names: Erbitux
  Arms: LY3537982 (Dose Expansion); LY3537982 (Dose Optimization)
Drug: Pemetrexed — Intravenous
  Other Names: LY231514; Alimta
  Arms: LY3537982 (Dose Expansion)
Drug: Cisplatin — Intravenous
  Arms: LY3537982 (Dose Expansion)
Drug: Carboplatin — Intravenous
  Arms: LY3537982 (Dose Expansion)

SUMMARY:
The purpose of this study is to find out whether the study drug, LY3537982, is safe and effective in cancer patients who have a specific genetic mutation (KRAS G12C). Patients must have already received or were not able to tolerate the standard of care, except for specific groups who have not had cancer treatment. The study will last up to approximately 4 years.

DETAILED DESCRIPTION:
This is an open-label, multicenter Phase 1/2 study to evaluate safety, tolerability, and preliminary efficacy of oral LY3537982 in patients with KRAS G12C-mutant solid tumors.

This study will be conducted in 4 parts: Phase 1a dose escalation, Phase 1b dose expansion, Phase 1b dose optimization, and Phase 2. KRAS G12C mutations will be identified through standard of care testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients have measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
* Patients must have disease with evidence of KRAS G12C mutation in tumor tissue or circulating tumor deoxyribonucleic acid (DNA).
* Participants must have a histological or a cytologically proven diagnosis of locally advanced, unresectable, and/or metastatic cancer and meet cohort-specific criteria.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Have adequate organ function.
* Have discontinued all previous treatments for cancer with resolution of any significant ongoing adverse events (AEs), (except in certain scenarios).
* Must be able to swallow capsule/tablet.
* Agree and adhere to contraceptive use, if applicable.
* For some parts of the study, (i.e., one of the two arms with LY3537982 in combination with pembrolizumab and the arm of LY3537982 in combination with pembrolizumab, pemetrexed, and platinum therapy) histologically or cytologically confirmed Stage IIIB-IIIC or Stage IV NSCLC that is previously untreated in the advanced/metastatic setting and not suitable for curative intent radical surgery or radiation therapy. Previously untreated patients who received adjuvant and neoadjuvant therapy are eligible if the last dose of the systemic treatment was completed at least 6 months prior to enrollment. For untreated patients in the arm with LY3537982 in combination with pembrolizumab noted above, a single cycle of pembrolizumab may be initiated within 21 days prior to enrollment. For untreated patients in the arm of LY3537982 in combination with pembrolizumab, pemetrexed, and platinum therapy, a single cycle of any or all of the drugs other than LY3537982 may be initiated within 21 days prior to enrollment. Start of study treatment may be delayed to allow sufficient time for recovery from treatment-related toxicity.
* For one part of the study, participants must have received at least one prior oxaliplatin- or irinotecan-containing regimen for advanced or metastatic CRC.

Exclusion Criteria:

* Disease suitable for local therapy administered with curative intent.
* Have an active, ongoing, or untreated infection.
* Have a serious pre-existing medical condition(s) that, in the judgment of the investigator, would preclude participation in this study.
* Have a serious cardiac condition.
* Have a second active primary malignancy or have been diagnosed and/or treated for an additional malignancy within 3 years prior to enrollment.
* For some parts of the study only: have untreated active central nervous system (CNS) metastases and/or leptomeningeal disease. Patients with treated CNS metastases are eligible for this study if their disease is asymptomatic, radiographically stable for at least 30 days, and they do not require treatment with steroids in the two-week period prior to study treatment. Patients with active CNS metastases are eligible for one part of the study.
* Have received prior treatment with any KRAS G12C small molecule inhibitor, except in certain scenarios where such prior therapy is allowed as per protocol.
* The following patients will be excluded from some parts of the study:

  * Experienced certain serious side effects with prior immunotherapy.
  * Have an active autoimmune disease that has required systemic anti-autoimmune treatment in the past 2 years.
  * Have received a live vaccine within 30 days prior to the first dose of study drug.
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial through 35 days after the last dose of study medication.
* Known allergic reaction against any of the components of the study treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: To determine the recommended phase 2 dose (RP2D) of LY3537982 monotherapy | Cycle 1 (21 Days)
  Measured by the number of patients with dose-limiting toxicities (DLTs)
Phase 1b: To assess the safety and tolerability of LY3537982 when administered alone or in combination with other investigational agents | Cycle 1 (21 Days)
  Measured by the number of patients with dose-limiting toxicities (DLTs)
Phase 1b: To determine the optimal dose of LY3537982 to be administered to treatment-naïve participants with advanced NSCLC in combination with pembrolizumab | Estimated up to 2 years
  Measured by TEAEs
To determine the optimal dose of LY3537982 to be administered to participants who have received at least one prior oxaliplatin- or irinotecan-containing regimen for advanced or metastatic CRC in combination with cetuximab | Estimated up to 2 years
To assess the antitumor activity of LY3537982 monotherapy in participants with advanced pancreatic cancer with KRAS G12C mutation | Estimated up to 2 years

SECONDARY OUTCOMES:
To assess preliminary antitumor activity of LY3537982 when administered alone or in combination with other investigational agents: Objective response rate (ORR) | Estimated up to 2 years
  ORR
To assess the preliminary antitumor activity of LY3537982 when administered alone or in combination with other investigational agents: Duration of Response (DOR) | Estimated up to 2 years
  DOR
To assess the preliminary antitumor activity of LY3537982 when administered alone or in combination with other investigational agents: Best Overall Response (BOR) | Estimated up to 2 years
  BOR
To assess the preliminary antitumor activity of LY3537982 when administered alone or in combination with other investigational agents: Time to response (TTR) | Estimated up to 2 years
  TTR
To assess the preliminary antitumor activity of LY3537982 when administered alone or in combination with other investigational agents: Disease control rate (DCR) | Estimated up to 2 years
  DCR
To assess the preliminary antitumor activity of LY3537982 when administered alone or in combination with other investigational agents: Progression-free survival (PFS) | Estimated up to 2 years
  PFS
To assess the preliminary antitumor activity of LY3537982 when administered alone or in combination with other investigational agents: Overall survival (OS) | Estimated up to 2 years
  OS
To assess the preliminary antitumor activity of LY3537982 when administered alone or in combination with other investigational agents: Intracranial DOR based on modified RECIST v1.1 (Certain arms of the study only) | Estimated up to 2 years
  Intracranial DOR
To assess the preliminary antitumor activity of LY3537982 when administered alone or in combination with other investigational agents: Whole-body ORR based on RECIST v1.1 and modified RECIST v1.1 (Certain arms of the study only) | Estimated up to 2 years
  Whole-body ORR
To characterize the pharmacokinetics (PK) properties of LY3537982: Area under the plasma concentration versus time curve (AUC) | Predose estimated up to 2 years
  PK: AUC of LY3537982
To characterize the PK properties of LY3537982: Maximum drug concentration (Cmax) | Predose estimated up to 2 years
  PK: Cmax of LY3537982

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - USC Norris Cancer Hospital, Los Angeles, California
  - Chao Family Comprehensive Cancer Ctr., Orange, California
  - Yale-New Haven Hospital, New Haven, Connecticut
  - AdventHealth Orlando, Orlando, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Indiana Univ Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Health Network, Indianapolis, Indiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Health- Long Island, Mineola, New York
  - NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Cancer Institute - Elizabeth, Charlotte, North Carolina
  - Novant Health Cancer Institute - Forsyth, Winston-Salem, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Vanderbilt Univeristy School of Medicine, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - Inova Health System IRB, Fairfax, Virginia
  - USO-Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Wisconsin-Madison Hospital and Health Clinic, Madison, Wisconsin
- Australia (5):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Cancer Research SA, Adelaide, South Australia
  - Peninsula and Southeast Oncology, Frankston, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hospital (Ontario), Toronto, Ontario
- France (5):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Institut du Cancer de Montpellier - Val d'aurelle, Montpellier
  - Institut Claudius Regaud - IUCT Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Japan (6):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeonranamdo
  - Seoul National University Hospital, Seoul, Korea
  - Asan Medical Center, Seoul, Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study of LY3537982 in Cancer Patients with a Specific Genetic Mutation (KRAS G12C) — https://trials.lilly.com/en-US/trial/295242